CLINICAL TRIAL: NCT04700501
Title: On-line Cognitive Behavioural Therapy Intervention in Pregnancy 'Enjoy Your Bump': an Antenatal Intervention for Perinatal Anxiety
Brief Title: Enjoy Your Bump - Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Tommy's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AC20128; 285587 (Other: IRAS); 20/SS/0100 (Other: Reviewing Ethics Committee (REC))
Record Dates: First submitted 2020-11-30; First posted 2021-01-08 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2021-09

CONDITIONS: Antenatal Depression

STUDY DESIGN:
Intervention Model Description: implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EYB Implementation study (Other): All participants will have the opportunity to access an online CBT life skills learning programme.
  Interventions: Other: Enjoy Your Bump - CBT life skills learning programme

INTERVENTIONS:
Other: Enjoy Your Bump - CBT life skills learning programme — Antenatal use of an online Cognitive Behavioural Therapy life skills learning programme to improve maternal feelings of anxiety and low mood.

SUMMARY:
Enjoy Your Bump is an implementation study relating to antenatal maternal mental health in women who have mild to moderate feelings of depression and anxiety. The investigators aim to address the following research question: Is a pregnancy-specific online CBT based life skills course (EYB) delivered antenatally clinically effective in improving maternal anxiety symptom scores immediately post-intervention and at 12 weeks postpartum?

The investigators hypothesise that a pregnancy specific on-line CBT intervention delivered antenatally will improve PNMH during pregnancy and that this will be sustained at 3 months post-partum with beneficial effects for mother and child.

The pregnancy specific online CBT tool Enjoy Your Bump (EYB) course teaches CBT-based life skills to expecting mothers in a fun and low-jargon way. Participants are asked to complete 5 'core' modules and encouraged to take their time to learn, reflect and practice these new life skills.

The investigators anticipate recruiting approximately 100 women to participate in this implementation study. Mental health assessments will be conducted before starting the CBT programme, on completion of the programme and again at 6-12 weeks postnatal. The investigators anticipate an improvement in maternal mental health assessment scores in women who have completed the course and the investigators hope to observe a longer term effect in scores at 6-12 weeks postnatal.

DETAILED DESCRIPTION:
One in four women have mental health problems, such as feeling anxious or depressed, during pregnancy and following childbirth. This not only impacts on the woman's own wellbeing but can also adversely affect the physical development and mental wellbeing of her child. The National Health Service (NHS) Long Term Plan aims to be able to provide better access to quality psychological interventions for women with mental health problems in pregnancy. Since the start of the Covid-19 outbreak in March 2020, pregnant women have been placed in a vulnerable group. There have been dramatic changes to maternity services in the community and hospital settings with remote midwife visits and changes to antenatal services. The normal support from friends and family has been reduced due to the current social distancing guidelines. This has all led to an increase in levels of stress and anxiety in the antenatal population.

The investigators have developed a unique pregnancy-specific on-line educational CBT based life skills course called Enjoy Your Bump (EYB). Unlike other CBT tools currently in use, this tool is specifically designed for use by pregnant women with chronic PNMH problems like elevated anxiety, mild depressive symptoms or high levels of self-reported stress. It also addresses specific concerns that women have during pregnancy, is the only pregnancy specific on-line CBT tool available and teaches CBT-based life skills in a fun and low-jargon way.

This implementation study will be open to any pregnant women in NHS Lothian who are experiencing mild or moderate symptoms of anxiety or depression. All pregnant women have access to an antenatal booking appointment with the community midwife following a positive pregnancy test. Women receive routine antenatal appointments during other stages of pregnancy and can participate in the study at any time point up to 32 weeks of pregnancy. During the booking appointment women are routinely asked two mental health questions:

1. During the past month has the participant often been bothered by feeling down, depressed or hopeless?"
2. During the past month has the participant often been bothered by having little interest or pleasure in doing things?"

If participants answer yes to either of these questions, the midwife can direct them to the online Enjoy Your Bump study website to gain further information about the study.

Information about this study will also be displayed in maternity waiting rooms in hospitals and on-line websites and women can self refer to participate.

Following completion of three baseline questionnaires, the participants will be provided with a link to the Enjoy Your Bump website. It can be completed using a tablet, smart phone, computer or kindle and is delivered as a modular intervention.

Women are asked to complete 5 'core' modules. There are additional optional modules and support materials the women can access to support their journey through the programme. The modules are supported by completion of 'worksheets' which can be accessed electronically. EYB is unique, as it is tailored to include specific issues relevant to pregnancy. At approximately 36 weeks gestation (after completion of the modules) the participants will be asked to complete 3 short questionnaires either by phone or by an email link to the study website. As part of routine practice all women receive a 6-12 week community follow up appointment by a health care professional. During this appointment the EPDS questionnaire is collected to assess postnatal mental Health.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or over,
* Capacity to give informed consent to participate in the study,
* Mild to moderate chronic Perinatal mental health (PMH) problems Score ≥3 on PHQ- 2,
* 8-32 week gestation

Exclusion Criteria:

* Severe Perinatal mental health problem - schizophrenia, bipolar disorder,
* Substance abuse/dependence,
* Active risk of self-harm,
* Insufficient English language to engage with intervention,
* No access to the internet

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
To measure any change from baseline mental health scores when the General Anxiety Disorder-7 (GAD-7) is repeated on completion of the course, or at 36 weeks' gestation. | Through study completion, up to 1 year
  To determine if a pregnancy-specific online Cognitive Behavioural Therapy (CBT) based life skills course delivered antenatally is effective in improving short term maternal mental health scores following the CBT intervention. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
To measure any change from baseline mental health scores when the Patient Health Questionnaire -8 (PHQ-8) is repeated on completion of the course, or at 36 weeks' gestation. | Through study completion, up to 1 year
  To determine if a pregnancy-specific online Cognitive Behavioural Therapy (CBT) based life skills course delivered antenatally is effective in improving short term maternal mental health scores following the CBT intervention. Eight patient questions, each of which is scored 0 to 3, providing a 0 to 24 severity score. This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of - not at all, several days, more than half the days, and nearly every day, respectively. PHQ-8 total score for the eight items ranges from 0 to 24. Scores of 5, 10, 15, and 20 represent cut off points for mild, moderate, moderately severe and severe depression, respectively.
To measure any change from baseline mental health scores when the Edinburgh Postnatal Depression Score is repeated on completion of the course, or at 36 weeks' gestation. | Through study completion, up to 1 year
  To determine if a pregnancy-specific online Cognitive Behavioural Therapy (CBT) based life skills course delivered antenatally is effective in improving short term maternal mental health scores following the CBT intervention. The scale consists of 10 short statements. A mother checks off one of four possible answers that is closest to how she has felt during the past week. Responses are scored 0, 1, 2 and 3 based on the seriousness of the symptom. The total score is found by adding together the scores for each of the 10 items. None or minimal depression (0-6), Mild depression (7-13), Moderate depression (14-19), Severe depression (19-30).

SECONDARY OUTCOMES:
To measure the post-natal Edinburgh Postnatal Depression Scale (EPDS) scores when taken at 6-12 weeks by NHS Health Visitors. | Through study completion, up to 1 year
  To determine if a pregnancy-specific online Cognitive Behavioural Therapy (CBT) based life skills course delivered antenatally is effective in improving maternal mental health scores at 6- 12 weeks following birth. The scale consists of 10 short statements. A mother checks off one of four possible answers that is closest to how she has felt during the past week. Responses are scored 0, 1, 2 and 3 based on the seriousness of the symptom. The total score is found by adding together the scores for each of the 10 items. None or minimal depression (0-6), Mild depression (7-13), Moderate depression (14-19), Severe depression (19-30). A higher score is indicative of poorer mental health.
To measure the number of participants consented into the study. | Through study completion, up to 1 year
  To assess the uptake and completion of the CBT course.

CONTACTS AND LOCATIONS:
Overall Officials: Professor R Reynolds, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Queens Medical Research Facility, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antenatal and postnatal mental health: clinical management and service guidance. National Institute of Health and Clinical Excellence (NICE) guidelines [CG192] Published date: December 2014
- [Background] Saving Lives, Improving Mothers' Care. Lessons learned to inform future maternity care from the UK and Ireland Confidential Enquiries into Maternal Deaths and Morbidity 2009-2012
- [Background] Bauer A, Parsonage M, Knapp M, Lemmi V, Adelaja B. The costs of perinatal mental health problems. London School of Economics and Political Science. 2014.
- [Background] Heron J, O'Connor TG, Evans J, Golding J, Glover V; ALSPAC Study Team. The course of anxiety and depression through pregnancy and the postpartum in a community sample. J Affect Disord. 2004 May;80(1):65-73. doi: 10.1016/j.jad.2003.08.004. PMID 15094259
- [Background] Evans J, Heron J, Francomb H, Oke S, Golding J. Cohort study of depressed mood during pregnancy and after childbirth. BMJ. 2001 Aug 4;323(7307):257-60. doi: 10.1136/bmj.323.7307.257. PMID 11485953
- [Background] Ashford MT, Olander EK, Ayers S. Computer- or web-based interventions for perinatal mental health: A systematic review. J Affect Disord. 2016 Jun;197:134-46. doi: 10.1016/j.jad.2016.02.057. Epub 2016 Mar 9. PMID 26991368
- [Background] Lee EW, Denison FC, Hor K, Reynolds RM. Web-based interventions for prevention and treatment of perinatal mood disorders: a systematic review. BMC Pregnancy Childbirth. 2016 Feb 29;16:38. doi: 10.1186/s12884-016-0831-1. PMID 26928898
- See also: Chief Medical Office Annual Report 2014: women's health — https://www.gov.uk/government/publications/chief-medical-officer-annual-report-2014-womens-health
- See also: Perinatal mental health services needs assessment and recommendations. — https://www.gov.scot/publications/delivering-effective-services-needs-assessment-service-recommendations-specialist-universal-perinatal-mental-health-services/
- See also: Maternal mental health alliance — https://maternalmentalhealthalliance.org/
- See also: Five year forward view for mental health. one year on — https://www.england.nhs.uk/publication/five-year-forward-view-for-mental-health-one-year-on-report/